CLINICAL TRIAL: NCT05256732
Title: Phase 1, Multiple Dose, Randomized, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of AT-527 Following Oral Administration Under Fasting Conditions or With a Meal in Healthy Adult Subjects
Brief Title: Study of AT-527 in Healthy Subjects Under Fasting Conditions or With a Meal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AT-03A-015
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Healthy Volunteer Study
MeSH Terms: interventions — AT-511

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- AT-527 (Experimental)
  Interventions: Drug: AT-527 fasted; Drug: AT-527 fed
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo Comparator fasted; Other: Placebo Comparator fed
- AT-527 BID (Experimental)
  Interventions: Drug: AT-527
- AT-527 single dose fasted/fed (Experimental)
  Interventions: Drug: AT-527 single dose

INTERVENTIONS:
Drug: AT-527 fasted — AT-527 administered twice daily (BID) for 5 days fasted
  Other Names: Bemnifosbuvir
  Arms: AT-527
Other: Placebo Comparator fasted — Matching placebo administered twice daily (BID) for 5 days fasted
  Arms: Placebo
Drug: AT-527 fed — AT-527 administered twice daily (BID) for 5 days fed
  Other Names: Bemnifosbuvir
  Arms: AT-527
Other: Placebo Comparator fed — Matching placebo administered twice daily (BID) for 5 days fed
  Arms: Placebo
Drug: AT-527 — AT-527 administered twice daily (BID)
  Other Names: Bemnifosbuvir
  Arms: AT-527 BID
Drug: AT-527 single dose — AT-527 single dose fasted/fed cross-over
  Other Names: Bemnifosbuvir
  Arms: AT-527 single dose fasted/fed

SUMMARY:
This study will assess the safety, tolerability and pharmacokinetics (PK) of AT-527 following oral administration under fasting conditions or with a meal in healthy adult subjects

ELIGIBILITY:
Inclusion Criteria:

* Must agree to use two methods of birth control from Screening through 90 days after administration of the last dose of study drug
* Females must have a negative pregnancy test at Screening and prior to dosing
* Minimum body weight of 50 kg and body mass index (BMI) of 18-32 kg/m2
* Willing to comply with the study requirements and to provide written informed consent

Exclusion Criteria:

* Pregnant or breastfeeding
* Infected with hepatitis B virus, hepatitis C virus, HIV or COVID-19
* Abuse of alcohol or drugs
* Use of other investigational drugs within 28 days of dosing
* Other clinically significant medical conditions or laboratory abnormalities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of AT-527 | Day 1
  Maximum plasma concentration (Cmax)
Pharmacokinetics (PK) of AT-527 | Day 1
  Area under the concentration-time curve (AUC)
Pharmacokinetics (PK) of AT-527 | Day 1
  Trough plasma concentration (Ctrough)
Proportions of subjects experiencing treatment-emergent adverse events | Day 1-10

CONTACTS AND LOCATIONS:
Locations (1):
- Atea Study Site, Québec, Montreal, Quebec, Canada